CLINICAL TRIAL: NCT00460265
Title: A Phase 3 Randomized Trial of Chemotherapy With or Without Panitumumab in Patients With Metastatic and/or Recurrent Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Study of Panitumumab Efficacy in Patients With Recurrent and/or Metastatic Head and Neck Cancer
Acronym: SPECTRUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050251
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Recurrent and/or Metastatic Head and Neck Cancer
Keywords: Squamous Cell Carcinoma; Epidermal Growth Factor; Epidermal Growth Factor Receptor; SCCHN; Metastatic Head and Neck Cancer; EGFr; Head and Neck Cancer; Recurrent Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM 2 (Active Comparator): Arm 2 consists of Cisplatin and 5-FU
  Interventions: Drug: ARM 2
- ARM 1 (Experimental): ARM 1 Consists of Panitumumab plus Cisplatin and 5-FU
  Interventions: Drug: ARM 1

INTERVENTIONS:
Drug: ARM 2 — Subjects will receive Cisplatin plus 5FU
  Arms: ARM 2
Drug: ARM 1 — Subjects will receive Panitumumab plus cisplatin and 5FU
  Arms: ARM 1

SUMMARY:
The purpose of this study is to determine the treatment effect of Panitumumab in combination with chemotherapy versus chemotherapy alone as first line therapy for metastatic and/or recurrent squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman at least 18 years old.
* Histologically or cytologically confirmed metastatic and/or recurrent squamous cell carcinoma (or its variants) of the head and neck.
* Diagnosis of metastatic disease and/or recurrent disease following locoregional therapy and determined to be incurable by surgery or radiotherapy.
* Subjects who have received radiation as primary therapy are eligible if locoregional recurrence is in the field of radiation and has occurred ≥6 months after the completion of radiation therapy. Subjects whose locoregional recurrence is solely outside the field of radiation are eligible if the recurrence has occurred ≥ 3 months after the completion of radiation therapy.
* Measurable and non-measurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* History or known presence of Central Nervous System (CNS) metastases.
* History of another primary cancer, except: curatively treated in situ cervical cancer, or curatively resected non-melanoma skin cancer, or other primary solid tumor curatively treated with no known active disease present and no treatment administered for ≥ 2 years before randomization.
* Nasopharyngeal carcinoma.
* Prior systemic treatment for metastatic and/or recurrent SCCHN
* Prior cisplatin containing induction chemotherapy followed by cisplatin containing chemoradiotherapy
* Prior anti-EGFr (Epidermal growth factor receptor) antibody therapy or treatment with small molecule EGFr inhibitors
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) less than or equal to 1 year prior to randomization. History of interstitial lung disease (eg, pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest computerized tomography (CT) scan.
* Symptomatic peripheral neuropathy grade ≥ 2 based on the CTCAE v3.0
* Grade ≥ 3 hearing loss based on the Common Terminology Criteria for Adverse Events (CTCAE) v3.0 Auditory/Ear (Hearing [without monitoring program])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2007-05; Primary Completion 2010-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Bach B, et al.SPECTRUM biomarkers HPV.Journal-004521;
- [Background] Vermorken JB, Stohlmacher-Williams J, Davidenko I, Licitra L, Winquist E, Villanueva C, Foa P, Rottey S, Skladowski K, Tahara M, Pai VR, Faivre S, Blajman CR, Forastiere AA, Stein BN, Oliner KS, Pan Z, Bach BA; SPECTRUM investigators. Cisplatin and fluorouracil with or without panitumumab in patients with recurrent or metastatic squamous-cell carcinoma of the head and neck (SPECTRUM): an open-label phase 3 randomised trial. Lancet Oncol. 2013 Jul;14(8):697-710. doi: 10.1016/S1470-2045(13)70181-5. Epub 2013 Jun 6. PMID 23746666
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 25 May 2007 to 10 March 2009.
Groups:
- Panitumumab Plus Chemotherapy: Consists of Panitumumab plus Cisplatin and 5-FU
- Chemotherapy Alone: Consists of Cisplatin and 5-FU
Period: Overall Study
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Started | 328 | 330
Randomized While Alive | 327 (1 subject was randomized by error after death) | 330
Received Study Medication | 325 | 325
Completed | 243 (Completed study=death) | 241 (Completed study=death)
Not Completed | 85 | 89
Not completed — Lost to Follow-up | 14 | 15
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 10 | 25
Not completed — Ongoing | 60 | 47

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone | Total
Number analyzed (Participants) | 327 | 330 | 657
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (8.5) | 58.6 (7.8) | 58.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 87
  Male | 283 | 287 | 570
Race/Ethnicity, Customized [Number; unit: subjects]
  White or Caucasian | 268 | 271 | 539
  Black or African American | 4 | 2 | 6
  Hispanic or Latino | 13 | 12 | 25
  Asian | 25 | 30 | 55
  Japanese | 13 | 7 | 20
  Aborigine | 1 | 0 | 1
  Other | 3 | 6 | 9
  Unknown/Missing | 0 | 2 | 2
Previously treated with chemotherapy and/or radiotherapy, Yes/No [Number; unit: subjects]
  Yes | 267 | 263 | 530
  No | 60 | 67 | 127
ECOG perfomance score, 0/1/2 [Number; unit: subjects]
  0 | 98 | 98 | 196
  1 | 227 | 228 | 455
  2 | 2 | 4 | 6
Primary tumor site, oropharynx&larynx/oral cavity&hypopharynx [Number; unit: subjects]
  Oropharynx and larynx | 186 | 191 | 377
  Oral cavity and hypopharynx | 141 | 139 | 280

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from randomization to death
Time Frame: Upto 56 months
Population: Intention to treat (ITT)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 327 | 330
months | 11.1 [9.8 to 12.2] | 9.0 [8.1 to 11.2]
Statistical Analysis 1: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; p = 0.1403, Log Rank; Stratified by IVRS randomization factors (ECOG(0:1),previously treated w/ CT/RT(yes:no),primary tumor site(oropharynx/larynx:oral cavity/hypopharynx)); Hazard Ratio (HR) = 0.873, 95% CI [0.729 to 1.046] — Hazard ratio from Cox proportional hazards model stratified by IVRS randomization factors; hazard ratio presented as panitumumab plus chemotherapy:chemotherapy alone

2. Secondary Outcome: Overall Response Rate
Description: An objective tumor response of complete or partial response per modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.0 that was confirmed no less than 28 days after the criteria for response were first met. Complete response = disappearance of all target lesions and partial response = ≥30% reduction in lesion size.
Time Frame: Every 6 weeks until disease progression, up to 56 months
Population: The subset of subjects in the ITT analysis set with at least one baseline uni-dimensionally measurable lesion using a modified version of the RECIST v1.0 (see protocol Appendix H)
Measure: Number; unit: subjects
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 278 | 288
subjects | 101 | 73
Statistical Analysis 1: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; Difference in percentages = 10.98, 95% CI [3.13 to 18.68]
Statistical Analysis 2: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; Odds Ratio (OR) = 1.69, 95% CI [1.15 to 2.44]

3. Secondary Outcome: Duration of Response
Description: Time from the first confirmed objective response of complete or partial response (that is subsequently confirmed at least 28 days later) to disease progression using a modified version of the RECIST v1.0 (see protocol Appendix H).
Time Frame: Every 6 weeks until disease progression, up to 56 months
Population: Included only those subjects with a confirmed complete or partial response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 101 | 73
months | 5.6 [4.8 to 6.2] | 5.7 [4.7 to 6.2]

4. Secondary Outcome: Time to Progression
Description: Time from randomization date to date of disease progression using a modified version of the RECIST 1.0 (see protocol Appendix H)
Time Frame: Every 6 weeks until disease progression, up to 56 months
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 327 | 330
months | 6.8 [5.9 to 6.9] | 5.6 [5.2 to 5.8]

5. Secondary Outcome: Time to Response
Description: Time from randomization date to the first confirmed objective response of complete or partial response (that is subsequently confirmed at least 28 days later) using a modified version of the RECIST v1.0.
Time Frame: Every 6 weeks until disease progression, upto 56 months
Population: Included only those subjects with a confirmed complete response or partial response.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 101 | 73
months | 1.4 [1.3 to 2.5] | 1.5 [1.3 to 2.6]

6. Secondary Outcome: Progression Free Survival
Description: Time from randomization date to date of disease progression using a modified version of the RECIST v1.0 or death.
Time Frame: Every 6 weeks until disease progression or deaths, upto 56 months
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 327 | 330
months | 5.8 [5.6 to 6.6] | 4.6 [4.1 to 5.4]
Statistical Analysis 1: Comparison: Panitumumab Plus Chemotherapy vs Chemotherapy Alone; Test type: Superiority or Other; Hazard Ratio (HR) = 0.780, 95% CI [0.659 to 0.922] — Cox proportional hazards model stratified by IVRS randomization factors

ADVERSE EVENTS:
Time Frame: The day of the first dose of study therapy through 33 days since the last dose date (up to 56 months)
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Panitumumab Plus Chemotherapy | Chemotherapy Alone
Serious Adverse Events (participants affected / at risk) | 157/325 | 139/325
Other Adverse Events (participants affected / at risk) | 311/325 | 301/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus Chemotherapy (N=325) | Chemotherapy Alone (N=325)
Anaemia (Blood and lymphatic system disorders) | 15 | 16
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 18 | 12
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 11 | 14
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 4
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 4
Cardiac failure (Cardiac disorders) | 3 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 5
Cardiopulmonary failure (Cardiac disorders) | 2 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ichthyosis (Congenital, familial and genetic disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2
Papilloedema (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Aphagia (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 4
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 7
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 2
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 6
Necrotising colitis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 8
Abasia (General disorders) | 0 | 1
Asthenia (General disorders) | 8 | 3
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 2 | 2
Device occlusion (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 1
General physical health deterioration (General disorders) | 10 | 9
Hyperpyrexia (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Medical device complication (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 5 | 7
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 5 | 0
Pyrexia (General disorders) | 5 | 10
Sudden death (General disorders) | 1 | 2
Thrombosis in device (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Abscess (Infections and infestations) | 2 | 0
Abscess neck (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 1 | 0
Bronchiectasis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 2
Campylobacter infection (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 1
Clostridial infection (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 2 | 1
Erysipelas (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 2
Influenza (Infections and infestations) | 1 | 0
Laryngotracheitis obstructive (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 2
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Myiasis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 2 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pleural infection bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 10 | 13
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory moniliasis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 7 | 5
Septic shock (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal shock (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 4 | 1
White blood cell count decreased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 9
Dehydration (Metabolism and nutrition disorders) | 16 | 8
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 0
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3
Encephalopathy (Nervous system disorders) | 0 | 2
Epilepsy (Nervous system disorders) | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 2
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Radiculitis lumbosacral (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 5 | 5
Renal failure acute (Renal and urinary disorders) | 3 | 3
Renal impairment (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Anoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 0
Haemorrhage (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 7 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 0
Iliac artery embolism (Vascular disorders) | 1 | 0
Infarction (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus Chemotherapy (N=325) | Chemotherapy Alone (N=325)
Anaemia (Blood and lymphatic system disorders) | 132 | 126
Leukopenia (Blood and lymphatic system disorders) | 51 | 49
Neutropenia (Blood and lymphatic system disorders) | 157 | 140
Thrombocytopenia (Blood and lymphatic system disorders) | 74 | 74
Tinnitus (Ear and labyrinth disorders) | 21 | 28
Conjunctivitis (Eye disorders) | 23 | 4
Abdominal pain (Gastrointestinal disorders) | 20 | 10
Abdominal pain upper (Gastrointestinal disorders) | 22 | 18
Constipation (Gastrointestinal disorders) | 83 | 74
Diarrhoea (Gastrointestinal disorders) | 123 | 76
Dyspepsia (Gastrointestinal disorders) | 25 | 20
Dysphagia (Gastrointestinal disorders) | 23 | 24
Nausea (Gastrointestinal disorders) | 178 | 180
Stomatitis (Gastrointestinal disorders) | 67 | 62
Vomiting (Gastrointestinal disorders) | 140 | 126
Asthenia (General disorders) | 65 | 54
Fatigue (General disorders) | 90 | 81
Mucosal inflammation (General disorders) | 71 | 62
Oedema peripheral (General disorders) | 21 | 22
Pyrexia (General disorders) | 50 | 45
Paronychia (Infections and infestations) | 36 | 1
Blood creatinine increased (Investigations) | 23 | 33
Weight decreased (Investigations) | 81 | 54
Decreased appetite (Metabolism and nutrition disorders) | 94 | 90
Hypocalcaemia (Metabolism and nutrition disorders) | 42 | 20
Hypokalaemia (Metabolism and nutrition disorders) | 47 | 43
Hypomagnesaemia (Metabolism and nutrition disorders) | 132 | 66
Hyponatraemia (Metabolism and nutrition disorders) | 26 | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 15 | 20
Dizziness (Nervous system disorders) | 28 | 21
Headache (Nervous system disorders) | 29 | 35
Neuropathy peripheral (Nervous system disorders) | 27 | 20
Insomnia (Psychiatric disorders) | 27 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 19
Acne (Skin and subcutaneous tissue disorders) | 27 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 49 | 36
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 48 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 45 | 4
Erythema (Skin and subcutaneous tissue disorders) | 26 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 5
Rash (Skin and subcutaneous tissue disorders) | 165 | 9
Skin fissures (Skin and subcutaneous tissue disorders) | 24 | 0
Hypertension (Vascular disorders) | 16 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.